CLINICAL TRIAL: NCT01916473
Title: Epidural Versus Continuous Wound Ropivacaine Infusion: Effect on Acute and Chronic Pain After Myomectomy or Total Abdominal Hysterectomy. A Randomized Controlled Trial
Brief Title: Epidural Versus Continuous Wound Ropivacaine Infusion Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Argyro Fassoulaki, Professor of Anesthesiology, University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M-20/23-02-2010
Record Dates: First submitted 2013-07-15; First posted 2013-08-05 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Postoperative Analgesia
Keywords: Epidural analgesia; continuous wound infusion; ropivacaine; total abdominal hysterectomy
MeSH Terms: interventions — Analgesia, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epidural analgesia (Active Comparator): Epidural analgesia is provided with ropvacaine 0.2% given 6 hourly
  Interventions: Other: Epidural analgesia
- Continuous wound infusion (Experimental): The continuous wound infusion consists of 0.376% ropivacaine infusion in the wound area at a rate 2 ml per hour.
  Interventions: Other: Continuous wound infusion

INTERVENTIONS:
Other: Epidural analgesia — Epidural analgesia is provided with ropvacaine 0.2% given 6 hourly
  Arms: Epidural analgesia
Other: Continuous wound infusion — Continuous wound infusion via catheter
  Arms: Continuous wound infusion

SUMMARY:
Study Hypothesis: The analgesic requirements and pain scores postoperatively differ between the epidural and continuous wound infusion techniques.

DETAILED DESCRIPTION:
The analgesic requirements and pain scores postoperatively differ between the epidural and continuous wound infusion techniques, in patients undergoing myomectomy or hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

Patients ASA I-II scheduled for abdominal hysterectomy or myomectomy -

Exclusion Criteria:

Age older than 60 and younger than 25 years, body weight exceeding the 30% of the ideal, consumption of analgesics, sedatives, anxiolytics, antidepressants, calcium channel blockers, CNS disease or insulin dependent diabetes

-

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2010-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Postoperative morphine consumption | 2 hours postoperatively
Postoperative morphine consumption | 4 hours postoperatively
Postoperative morphine consumption | 8 hours postoperatively
Postoperative morphine consumption | 24 hours postoperatively
Postoperative morphine consumption | 48 hours postoperatively
Postoperative morphine consumption | 72 hours postoperatively
Postoperative morphine consumption | 3 months postoperatively
Postoperative morphine consumption | 6 months postoperatively

SECONDARY OUTCOMES:
pain scores | 2 hours postoperatively
pain scores | 4 hours postoperatively
pain scores | 8 hours postoperatively
pain scores | 24 hours postoperatively
pain scores | 48 hours postoperatively
pain scores | 72 hours postoperatively
pain scores | 3 months postoperatively
pain scores | 6 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Argyro Fassoulaki, MD,PhD, DEAA, Principal Investigator — University of Athens
Locations (1):
- Aretaieio Hospital, Athens, Greece